CLINICAL TRIAL: NCT03479216
Title: Comparison of Intra-articular Dexmedetomidine and Magnesium in Postoperative Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hande G. Aytuluk, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: U1111-1211-1791
Record Dates: First submitted 2018-03-21; First posted 2018-03-27 (Actual); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain; Intra-articular Injection; Dexmedetomidine; Magnesium Sulfate
Keywords: Analgesia; Anesthesia; Arthroscopy; Bupivacaine; Dexmedetomidine; Injections, Intra-Articular; Magnesium; Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dexmedetomidine; Bupivacaine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Precedex (Experimental): 5ml 0.25% Bupivacaine ve 50mcg Dexmetedomidin (diluted to 5ml with normal saline) intraarticularly at the end of surgery (total volume: 10 ml)
  Interventions: Drug: Precedex
- Magnesium Sulfate (Experimental): 5ml 0.25% Bupivacaine ve 5ml Magnesium Sulfate intraarticularly at the end of surgery (total volume: 10 ml)
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Precedex — 10 ml of Bupivacaine ve 50mcg Dexmetedomidin mixture will be injected intraarticularly at the end of the surgery.
  Other Names: bupivacaine
  Arms: Precedex
Drug: Magnesium Sulfate — 10 ml of Bupivacaine ve magnesium sulfate mixture will be injected intraarticularly at the end of the surgery.
  Other Names: bupivacaine
  Arms: Magnesium Sulfate

SUMMARY:
Arthroscopic meniscus surgeries are the most frequent orthopedic procedures. The objective of the study is to compare the effects of intraarticular local anesthetic and adjuvant (dexmedetomidine vs magnesium) combinations in postoperative pain and analgesic requirement. The investigators' hypothesis is adjuvants added to the local anesthetics decreases the total local anesthetic dose, provides more effective pain relief according to local anesthetic only, and decreases the postoperative systemic non-steroidal analgesic and opioid doses.

DETAILED DESCRIPTION:
Arthroscopic meniscus surgeries are the most frequent orthopedic procedures. However, irritation of free nerve endings in the synovial tissue and anterior fat pads and stretching and resection in the joint capsule lead to pain at various levels. Proper pain management enhances recovery, provides early mobilization and shortens length of hospital stay.

"Opioid-free" analgesia methods are frequently emphasized in published postoperative pain management guidelines and multimodal treatment approaches such as local anesthetic infiltration is recommended. In the treatment of knee pain, intra-articular drug injections are the most commonly used method because of minimal systemic side effects.

The drugs most commonly administered intraarticularly included local anesthetics (bupivacaine, levobupivacaine, lidocaine), opioids (morphine, fentanyl), magnesium sulfate, steroids, and α2 agonists (clonidine, dexmedetomidine).

Dexmedetomidine is a selective, specific, lipophilic and potent α2 adrenergic receptor agonist with sedative, anxiolytic, analgesic, antihypertensive and sympatholytic effects. It provides analgesic activity through both the central and peripheral nervous system. The analgesic effects of intra-articular administration of dexmedetomidine in arthroscopic surgeries have been demonstrated. Most side effects of this drug included hypotension and bradycardia. However, these side effects have never been encountered with intra-articular injection of the drug.

Magnesium is also an adjuvant drug which has a key role in nociceptive transmission, and acts as a NMDA (N-Methyl-D-Aspartate) antagonist in spinal neurons.

While opioid free anesthesia and analgesia methods gain importance nowadays, there has been increased interest in non-opioid analgesic drugs and multimodal analgesia applications. In order to increase the effects of local anesthetics and prolong their analgesic times, the addition of various adjuvants to local anesthetics is frequently used.

In the randomized controlled trials, intraarticular local anesthetic drugs combined with adjuvant drugs for postoperative analgesia were found to be superior to local anesthetic drugs alone. It is also known that local anesthetics have negative effects on chondrocytes. One of the goals of the investigators' in this study is to reduce the amount of local anesthetic used by adding adjuvant to local anesthetics.

In this study, the investigators plan to compare the efficacy of 2 adjuvants (magnesium sulfate and dexmedetomidine) combined with local anesthetics to be given intraarticularly for postoperative pain management after elective arthroscopic surgery.

Intraarticular high-volume drug injections may cause pain due to tension in the joint capsule. Additionally, the investigators aim to decrease the total drug volume with adjuvant drugs used in combination with local anesthetic, and thus to prevent joint capsule tension pain.

ELIGIBILITY:
Inclusion Criteria:

* age >18, <65
* scheduled for elective knee arthroscopy under spinal anesthesia
* ASA I and ASA II

Exclusion Criteria:

* age <18 and >65
* patients who received general anesthesia
* diabetes
* refusal of the patient
* known allergy to the specified drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tolga K Saracoglu, Ass Prof, Study Chair — Derince Training and Research Hospital
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
not decided yet

REFERENCES:
- [Result] Sun R, Zhao W, Hao Q, Tian H, Tian J, Li L, Jia W, Yang K. Intra-articular clonidine for post-operative analgesia following arthroscopic knee surgery: a systematic review and meta-analysis. Knee Surg Sports Traumatol Arthrosc. 2014 Sep;22(9):2076-84. doi: 10.1007/s00167-013-2615-8. Epub 2013 Jul 24. PMID 23881255
- [Result] Yang Y, Zeng C, Wei J, Li H, Yang T, Deng ZH, Li YS, Yang TB, Lei GH. Single-dose intra-articular bupivacaine plus morphine versus bupivacaine alone after arthroscopic knee surgery: a meta-analysis of randomized controlled trials. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):966-979. doi: 10.1007/s00167-015-3748-8. Epub 2015 Aug 12. PMID 26264382
- [Result] Gerlach AT, Dasta JF. Dexmedetomidine: an updated review. Ann Pharmacother. 2007 Feb;41(2):245-52. doi: 10.1345/aph.1H314. Epub 2007 Feb 13. Erratum In: Ann Pharmacother. 2007 Mar;41(3):530-1. PMID 17299013
- [Result] Alipour M, Tabari M, Faz RF, Makhmalbaf H, Salehi M, Moosavitekye SM. Effect of dexmedetomidine on postoperative pain in knee arthroscopic surgery; a randomized controlled clinical trial. Arch Bone Jt Surg. 2014 Mar;2(1):52-6. Epub 2014 Mar 15. PMID 25207314
- [Result] Li C, Qu J. Efficacy of dexmedetomidine for pain management in knee arthroscopy: A systematic review and meta-analysis. Medicine (Baltimore). 2017 Oct;96(43):e7938. doi: 10.1097/MD.0000000000007938. PMID 29068980
- [Result] Heydari SM, Hashemi SJ, Pourali S. The Comparison of Preventive Analgesic Effects of Ketamine, Paracetamol and Magnesium Sulfate on Postoperative Pain Control in Patients Undergoing Lower Limb Surgery: A Randomized Clinical Trial. Adv Biomed Res. 2017 Oct 25;6:134. doi: 10.4103/2277-9175.217217. eCollection 2017. PMID 29279832
- [Result] Kizilcik N, Ozler T, Menda F, Ulucay C, Koner O, Altintas F. The effects of intra-articular levobupivacain versus levobupivacain plus magnesium sulfate on postoperative analgesia in patients undergoing arthroscopic meniscectomy: A prospective randomized controlled study. Acta Orthop Traumatol Turc. 2017 Mar;51(2):104-109. doi: 10.1016/j.aott.2017.02.014. Epub 2017 Mar 15. PMID 28314555
- [Derived] Aytuluk HG, Gultekin A, Saracoglu KT. Comparison of intraarticular bupivacaine-dexmedetomidine and bupivacaine-magnesium sulfate for postoperative analgesia in arthroscopic meniscectomy: a randomized controlled clinical trial. Hippokratia. 2019 Apr-Jun;23(2):51-57. PMID 32265584

RESULTS

PARTICIPANT FLOW:
Recruitment Details: History of cardiac, hepatic or renal disorders, diabetes mellitus, chronic pain treatment, contraindication to/refusal of spinal anesthesia, a known allergy to the study drugs, or who refused to participate in the study were excluded.
  (10 patients excluded: 5 declined regional anesthesia, 4 had diabetes mellitus,1 failure of regional anesthesia)
Pre-assignment Details: 52 patients aged between 18 and 65 years with ASA I or II who were scheduled for elective arthroscopic meniscectomy under spinal anesthesia were included in this prospective, randomized, double-blind study.
Period: Overall Study
Arm/Group | Precedex | Magnesium Sulfate
Started | 31 | 31
Completed | 26 | 26
Not Completed | 5 | 5
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Physician Decision | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Precedex | Magnesium Sulfate | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Full Range); unit: years] | 41.62 [18 to 65] | 42.73 [23 to 59] | 42.18 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 20 | 22 | 42
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain
Description: postoperative pain scores (rest and movement) (ward) Pain scores were assessed with a 10-cm Visual Analogue Scale (VAS) (with 0 = no pain and 10 = the worst imaginable pain)
Time Frame: 24 hours
Population: visual analogue scale (VAS) scores at rest at 2nd hour (VAS2 R), 4th hour (VAS4 R), 6th hour (VAS6 R), 8th hour (VAS8 R), 12th hour (VAS12 R), 18th hour (VAS18 R) VAS scores at movement at 2nd hour (VAS2 M), 4th hour (VAS4 M), 6th hour (VAS6 M), 8th hour (VAS8 M), 12th hour (VAS12 M), 18th hour (VAS18 M)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Precedex | Magnesium Sulfate
Number analyzed (Participants) | 26 | 26
score on a scale
  VAS 2 R | 0 [0 to 0] | 0.04 [0 to 1]
  VAS2 M | 0.19 [0 to 2] | 0.23 [0 to 2]
  VAS4 R | 0.81 [0 to 3] | 0.12 [0 to 1]
  VAS4 M | 2.04 [0 to 6] | 1.19 [0 to 3]
  VAS6 R | 1.50 [0 to 4] | 1.31 [0 to 5]
  VAS6 M | 3.46 [0 to 8] | 3.31 [0 to 8]
  VAS8 R | 1.23 [0 to 5] | 1.77 [0 to 5]
  VAS8 M | 3.08 [0 to 8] | 4.08 [1 to 8]
  VAS12 R | 0.73 [0 to 5] | 1.15 [0 to 6]
  VAS12 M | 2.62 [0 to 6] | 3.19 [2 to 8]
  VAS18 R | 0.23 [0 to 1] | 0.27 [0 to 2]
  VAS18 M | 1.62 [0 to 4] | 1.69 [0 to 4]

2. Secondary Outcome: Postoperative Opioid/NSAID Consumption
Description: nonsteroid antiinflammatory drugs (NSAID) or opioid drugs that are applied to patients will be noted.
Time Frame: 24 hours
Measure: Number; unit: vials
Arm/Group | Precedex | Magnesium Sulfate
Number analyzed (Participants) | 26 | 26
vials
  NSAID | 17 | 14
  opioid | 0 | 1

3. Secondary Outcome: Rescue Analgesic Time
Description: Time to first analgesic demand at the orthopedics ward (from intraarticular injection to first analgesic requirement)
Time Frame: 24 hours
Population: Time to first analgesic demand at the orthopedics ward (from intra-articular injection to first analgesic requirement) was calculated in minutes among patients who required analgesics
Measure: Mean (Full Range); unit: minutes
Arm/Group | Precedex | Magnesium Sulfate
Number analyzed (Participants) | 15 | 13
minutes | 477.33 [240 to 840] | 498.46 [330 to 750]

4. Secondary Outcome: Surgery Time
Description: time from skin incision to closure
Time Frame: 24 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Precedex | Magnesium Sulfate
Number analyzed (Participants) | 26 | 26
minutes | 24.23 [15 to 35] | 25.58 [15 to 40]

5. Secondary Outcome: Time to the End of Spinal Anesthesia
Description: time from the start of spinal anesthesia (total block = Bromage 3) to the end of spinal anesthesia (Bromage 0)
Time Frame: 24 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Precedex | Magnesium Sulfate
Number analyzed (Participants) | 26 | 26
minutes | 148.1 [60 to 320] | 147.5 [70 to 300]

6. Secondary Outcome: Mobilization
Description: First mobilization time after surgery
Time Frame: 24 hours
Measure: Mean (Full Range); unit: minutes
Arm/Group | Precedex | Magnesium Sulfate
Number analyzed (Participants) | 26 | 26
minutes | 143.27 [75 to 300] | 139.42 [75 to 300]

7. Secondary Outcome: Number of Participants With Complications Due to Intraarticular Injection
Description: post-injection complications due to intraarticular injection will be noted.
Time Frame: 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Precedex | Magnesium Sulfate
Number analyzed (Participants) | 26 | 26
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: an average of 1 month (from hospitalization to re-admissions due to complications (if any))
Arm/Group | Precedex | Magnesium Sulfate
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-12): https://cdn.clinicaltrials.gov/large-docs/16/NCT03479216/Prot_SAP_000.pdf